CLINICAL TRIAL: NCT01556620
Title: The New 4 Wavelengths EQUANOX NIRS Sensor: Correlation and Detection of Ischemic Episodes. An Observational Comparative Study Versus PtiO2
Brief Title: Is NIRS Able to Detect Ischemia Following Brain Insult
Acronym: NIRS
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Principal Investigator, BORET Henry, Médecin en Chef, Direction Centrale du Service de Santé des Armées
Other Study IDs: DCSSA
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Brain Trauma; SAH; ICH
Keywords: PtiO2; NIRS
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We hypothesize that newly developped NIRS sensor (EQUANOX Advance™, 8004CA, NONIN Medical, USA)is able to detect ischemic events recorded by brain tissue oxygen probe (Licox, Integra Neurosciences, USA) and that values are correlated.

ELIGIBILITY:
Inclusion Criteria:

* Necessity of monitoring by PtiO2 and ICP

Exclusion Criteria:

* Inability to apply NIRS sensor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brain injury (head trauma, SAH, ICH)
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry BORET, MD, Principal Investigator — Direction Centrale du Service de Santé des Armées
Locations (1):
- Sainte Anne Military Teaching Hospital, Toulon, France